CLINICAL TRIAL: NCT03507530
Title: Investigating The Effects of Fear of Falling on Physical Performance and Quality of Life in Children With Duchenne Muscular Dystrophy
Brief Title: Effects of Fear of Falling on Physical Performance and Quality of Life in Children With Duchenne Muscular Dystrophy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Canan İpek (Other)
Responsible Party: Sponsor-Investigator, Canan İpek, Principal Investigator, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: GO 18/45
Record Dates: First submitted 2018-04-08; First posted 2018-04-25 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Neuromuscular Diseases; Duchenne Muscular Dystrophy; Dystrophy; Dystrophy, Muscular
Keywords: physiotherapy and rehabilitation; fear of falling; quality of life
MeSH Terms: conditions — Neuromuscular Diseases; Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessments — Falls related assessments, functional physical performance evaluations and quality of life assessments.

SUMMARY:
For ambulatory children with DMD, physiotherapy is aimed at protecting ambulation, improving motor performance to the best level and increasing quality of life. The investigators think that the treatment of children with Duchenne Muscular Dystrophy may become more effective with physiotherapy programs based on the comprehensive physiotherapy evaluation results, including the evaluation of fear of falling. This study investigates the fear of falling in children with Duchenne Muscular Dystrophy and questioning whether their fear of falling affects their quality of life and their physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Duchenne Muscular Dystrophy by a pediatric neurologist,
* Being volunteer,
* Being between 6 and 15 years old,
* Being between levels 1-5 according to the Brooke Lower Extremity Functional Classification developed to classify lower extremity functions in children with DMD,
* Being able to cooperate with the physiotherapist's directives.

Exclusion Criteria:

* Being between levels 6-10 (children who do not have independent ambulatory ability) according to the Brooke Lower Extremity Functional Classification,
* Not being able to cooperate with the physiotherapist's directives,
* End of the volunteering.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Duchenne Muscular Dystrophy, Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Pediatric Neuromuscular Diseases Unit.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Fear of Falling | 15-30 minutes
  "ICF Based 'Fear of Falling' Assessment in Pediatric Neuromuscular Diseases" is developed by researchers as examining the 'fear of falling' assessments in the literature and organizing the activities that children with Duchenne Muscular Dystrophy (DMD) may have experience fear of falling. There are six main titles which are based on DMD population and ICF headings. As follows: "Learning and Applying Knowledge", "General Tasks and Demands", "Mobility", "Self-Care", "Major Life Areas" and "Community, Social and Civic Living". It is a form total of 34 items which children with DMD answer to the fear of falling during different activities as "never = 0", "sometimes = 1", "always = 2" or "not applicable = NA". High scores indicate high fear of falling.

SECONDARY OUTCOMES:
History of Falls | 15-20 minutes
  Fall history of children with DMD is assessed using the 17-item History of Fall Questionnaire, which was developed by Ann Myers in 1996 and was later used to assess the fear of falling of individuals with Spinal Muscular Atrophy, a neuromuscular disease. Accordingly, past experiences of falling children are evaluated in sub-titles such as frequency, location, internal and external causes, injury.
Posture Analysis | 15-20 minutes
  Posture analysis is made by using "New York Posture Rating Scale".
Performance Evaluation | 6 minutes
  6 minute walking test (6MWT) are used.
Evaluation of Energy Consumption | 15-20 minutes
  Physiological Cost Index is used to evaluate energy consumption. It reflects the increased heart rate required for walking and is expressed as heartbeats per meter by formula: [Heart rate after 6MWT- Heart rate at rest]/Walking speed (m/min).
Fatigue | 15-20 minutes
  To evaluate the fatigue of the children with DMD, PedsQL Multidimensional Fatigue Scale is used. This scale assesses fatigue with a total of 18 items, 6 items in each of the 3 main headings: "General Fatigue", "Sleeping / Resting Fatigue" and "Cognitive Fatigue". There are three different forms for young children (5-7 years), children (8-12 years) and adolescents (13-17 years). All three forms have both child and parent reports. The reliability and validity of the scale is proven in Turkish.
Balance Assessment | 15-20 minutes
  The Pediatric Berg Balance Scale is used to assess the functional balance in the daily activities of children with DMD. The scale consists of 14 sections and each section is scored between 0-4; the highest score that can be taken from the scale is 56 and the higher scores show the better balance level.
Functional Walking Assessment | 5-10 minutes
  Gillette Functional Walking Scale is used for practical assessment of walking. The parent marks the item that best describes the child's ability to walk within 10 items. The high score means better walking ability.
Gait Analysis | 15-20 minutes
  Spatio-temporal characteristics of gait are assessed. Step length, stride length, step width (width of the walking base) and stance width are measured by footprint method which we use talcum powder to make them appear.The walking speed are recorded according to the 6MWT results.
Ambulation Assessment | 15-20 minutes
  The North Star Ambulatory Assessment which is a 17-item rating scale that is used to measure functional motor abilities in ambulant children with Duchenne Muscular Dystrophy (DMD) is used. The activities are scored as follows:
  2 - 'Normal' - no obvious modification of activity
  1 - Modified method but achieves goal independent of physical assistance from another 0 - Unable to achieve independently
Quality of Life | 15-20 minutes
  The Pediatric Outcomes Data Collection Instrument is used for a comprehensive assessment of quality of life of children with DMD. Functional dimensions are assessed include upper extremity functioning, transfers and basic mobility, sports and physical function, comfort/pain, global function (an average of the four previous scores), and happiness with physical condition. Scores for all dimensions are scaled from 0 to 100, with 100 being the highest level of function or happiness.
Activity Limitation | 5-10 minutes
  ACTIVLIM questionnaire is used which was designed to evaluate limitations in activities involving upper and lower limbs in adults and children with neuromuscular diseases, is linked to the domains of the Activities and Participation of the International Classification of Functioning, Disability and Health (ICF), and to its Children and Youth version (ICF-CY). There are 22 daily living activities and each item is answered on a 3-level scale (impossible, difficult, easy). The highest score that can be taken from the test is 44 and the higher scores indicate less activity limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No